CLINICAL TRIAL: NCT07345351
Title: Effects of Lifestyle Counseling Versus Lifestyle Counseling Combined With Clinical Pilates in Women With Temporomandibular Disorders
Brief Title: Lifestyle Counseling vs. Clinical Pilates in Women With Temporomandibular Disorders
Acronym: LiPi-TMD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Yasemin KARAASLAN, Principal Researcher, Head of Physiotherapy and Rehabilitation Department, Hatay Mustafa Kemal University, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBE2025-01
Record Dates: First submitted 2025-12-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Counseling; Health Counseling; Behavior Therapy
Keywords: Temporomandibular Disorders; Lifestyle Counseling; Clinical Pilates; Women's Health; Jaw Function; Functional Limitation
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Life Counselling (Active Comparator)
  Interventions: Behavioral: Life Counselling
- Arm 2: Life Counselling + Clinical Pilates (Experimental)
  Interventions: Behavioral: Life Counselling; Behavioral: Clinical Pilates

INTERVENTIONS:
Behavioral: Life Counselling — Participants receive individualized lifestyle counseling focused on stress management, physical activity, and sleep hygiene. Counseling sessions are conducted weekly for 8 weeks, delivered by a trained healthcare professional. The aim is to improve overall health behaviors related to temporomandibular disorder symptoms.
Behavioral: Clinical Pilates — Participants receive the same lifestyle counseling described above, combined with supervised clinical Pilates sessions. Pilates exercises focus on strengthening the core and improving posture and jaw function, conducted twice weekly for 8 weeks.
  Arms: Arm 2: Life Counselling + Clinical Pilates

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of lifestyle counseling alone compared to lifestyle counseling combined with Clinical Pilates in women with temporomandibular disorders (TMD). The study also aims to examine the effects of these interventions on pain, jaw function, posture, oral behaviors, psychological status, sleep quality, and quality of life.

The main questions this study aims to answer are:

Does adding Clinical Pilates to lifestyle counseling reduce pain levels in women with TMD more than lifestyle counseling alone?

Does the combined intervention improve jaw function, head posture, and oral behaviors?

What are the effects of these interventions on anxiety, sleep quality, and quality of life?

Researchers will compare lifestyle counseling alone with lifestyle counseling combined with a supervised Clinical Pilates program to determine whether the addition of Clinical Pilates provides greater clinical and psychosocial benefits.

Participants will be randomly assigned to one of two groups:

* Receive lifestyle counseling only (control group), or
* Participate in a supervised Clinical Pilates program twice weekly for 8 weeks in addition to lifestyle counseling (intervention group)

Undergo assessments at baseline (before any intervention) and after completion of the interventions.

Outcome measures will include assessments of pain, jaw function, posture, oral behaviors, psychological status, sleep quality, and quality of life.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental trial designed, which investigates the effectiveness of Clinical Pilates when added to lifestyle counseling, aims to contribute to the literature by evaluating its potential role in the treatment planning of women with TMD. Within the scope of this research, the therapeutic effects of Clinical Pilates will be examined.

The study will include agree to participate voluntarily, and meet the study criteria.

Inclusion criteria:

* Female participants aged between 18 and 45 years
* Diagnosed with temporomandibular disorder (according to DC/TMD diagnostic criteria)
* Experiencing TMD-related complaints for at least the past 3 months
* No prior experience with Pilates or lifestyle counseling
* No contraindications to exercise
* Diagnosed with muscle-related TMD

Exclusion Criteria:

* Presence of rheumatologic diseases
* Neurological disorders
* Pregnancy
* History of head or neck trauma
* Diagnosis of joint-related TMD (with or without reduction)

Participants will be randomly assigned into two groups:

* Group 1 (Control Group): Participants will receive lifestyle counseling only.
* Group 2 (Intervention Group): In addition to lifestyle counseling, participants will take part in a Clinical Pilates exercise program twice a week for a total duration of 8 weeks.

To evaluate the effects of the interventions, pre and post-treatment assessments will be conducted using the following outcome measures:

* Visual Analog Scale (VAS) and Graded Chronic Pain Scale Version 2.0 (GCPS v2.0) for pain assessment,
* Jaw Functional Limitation Scale-20 (JFLS-20) and Maximum Mouth Opening (MMO) for assessing jaw function,
* Craniovertebral Angle Measurement for evaluating head posture,
* Oral Behavior Checklist (OBC) for assessing oral parafunctions and bruxism,
* Generalized Anxiety Disorder-7 (GAD-7) for psychological status,
* Patient Health Questionnaire-15 (PHQ-15) for quality of life,
* Pittsburgh Sleep Quality Index (PSQI) for sleep quality.

Treatment Program Lifestyle counseling will be delivered as a structured program focusing on stress management, sleep hygiene, oral habits, and nutritional behaviors. Clinical Pilates exercises will be tailored to each participant's symptoms and supervised by an experienced physiotherapist. It will be elaborated during the reporting phase of the study and written into the article.

Sample size The sample size is a critical component in the study, and its consideration is essential for the interpretation of the results.

The sample size of the study will be determined using the GPower 3.1.9 software (GPower, Universität Düsseldorf, Germany) with a statistical power of 85% and a type I error rate of 5%. As there is no existing study with an effect size that precisely matches the current research design, the effect size obtained from a pilot study will be used, and a post-hoc power analysis will be conducted to finalize the sample size.

Statistical Analysis Descriptive statistics are reported as mean and standard deviation or median and mode. Categorical variables are defined with numbers and percentages. The normality assumption is tested using the Shapiro-Wilks test and graphs (hygtogram, QQ plot, etc.). When comparing two groups, the independent groups t-test is used if the assumptions are met, and the Mann-Whitney U test is used if the assumptions are not met. Two-way analysis of variance for repeated measures is used when the assumptions are met, and Friedman's test is used when the assumptions are not met. Chi-squared tests will be used to determine whether there is a significant difference between categorical variables. Analyses will be performed using IBM SPSS v.21 and the significance level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45
* Diagnosed with TMD (according to DC/TMD diagnostic criteria)
* Experiencing TMD symptoms for the past 3 months
* Have not previously received Pilates or lifestyle counseling
* Without any condition preventing exercise
* Diagnosed with muscle-related TMD

Exclusion Criteria:

* Rheumatological diseases
* Neurological disorders
* Pregnancy
* History of head or neck trauma
* Diagnosed with joint-related TMD (with or without reduction)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  Participants will be asked to mark their pain on a line ranging from 0 (no pain) to 10 (unbearable pain). Pain will be measured at rest and as palpation-induced pain (before and after palpation).
Graded Chronic Pain Scale Version 2.0 | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  The scale provides a simple, practical, and versatile assessment and is included in the DC/TMD diagnostic criteria. It consists of 8 questions: 3 questions assess pain intensity, 4 questions assess pain-related disability, and 1 question determines the number of painful days. For all questions except the 1st and 5th, participants are asked to rate their pain on a scale from 0 ("no pain") to 10 ("worst pain imaginable").
Jaw Functional Limitation Scale-20 | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  This is the most widely used self-report questionnaire for assessing jaw functional limitation in TMD. It is included among the recommended measures in the DC/TMD. The scale has three subscales evaluating masticatory function, jaw movements, and social/functional impact. It is scored using a 0-10 Likert scale. The Turkish version has proven reliability and validity (Yıldız, Kocaman, & Bingöl, 2024).
Maximum Mouth Opening | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  This is one of the objective indicators of functional limitation. A normal value is considered to be ≥40 mm. Participants will be asked to open their mouth as wide as possible, and the measurement will be taken using a caliper.
Craniovertebral Angle Measurement | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  This is a simple and clinically meaningful postural assessment method that provides information about head posture by measuring the forward position of the head. The angle between the line connecting the tragus (the prominence in front of the ear) and the C7 spinous process (lower part of the neck) and the horizontal plane is measured. A normal value is considered ≥48°. Values less than 48° are recorded as forward head posture (head anterior tilt) (Shaghayeghfard et al., 2016).
Oral Habits Checklist | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  Recommended in the DC/TMD protocol, this checklist is used to assess sleep and daytime bruxism as well as other parafunctional habits (e.g., pencil biting, nail biting) (Ohrbach & Dworkin, 2017).
Generalized Anxiety Disorder-7 Questionnaire (GAD-7) | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  This tool is used to screen for generalized anxiety disorder and measure the severity of general anxiety levels. It consists of 7 questions. Participants are asked how often they have experienced anxiety symptoms over the past two weeks. The scoring for each item is as follows: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day. The total score ranges from 0 to 21, with the following interpretations: 0-4 = Minimal anxiety, 5-9 = Mild anxiety, 10-14 = Moderate anxiety, and 15-21 = Severe anxiety (Konkan et al., 2013).
Patient Health Questionnaire-15 (PHQ-15) | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  Used to assess the frequency and severity of somatic (physical) symptoms and commonly applied for screening somatization disorder. Participants are asked how often they have experienced these symptoms over the past 4 weeks. The questionnaire includes 15 common physical symptoms (e.g., headache, stomach problems, fatigue, sleep disturbances). Each item is scored as 0 = Not at all, 1 = A little, and 2 = A lot. The total score ranges from 0 to 30, with the following interpretations: 0-4 = Low somatic symptom severity, 5-9 = Mild, 10-14 = Moderate, and 15 or higher = Severe somatic symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Each participant in the group will be evaluated twice. The first assessment will be conducted at the very beginning of the study before any intervention, and the second assessment will be performed after the interventions have been completed.
  Participants' sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The questionnaire consists of 24 items: 19 self-reported questions addressing factors related to sleep quality, and 5 items answered by a spouse or roommate. The 5 spouse/roommate items are clinically evaluated but not included in scoring. The 19 self-report items measure seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each question is scored from 0 to 3. The total PSQI score (ranging from 0 to 21) is calculated by summing the seven component scores. A total score of 5 or below indicates good sleep quality, while a score above 5 indicates poor sleep quality (Ağargün, Kara, & Anlar, 1996).

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Hatay, Turkey (Türkiye)